CLINICAL TRIAL: NCT01525017
Title: A Phase I Open-label Study to Evaluate Safety and Immunologic Response of COMBIG-DC Administered Intratumorally in Patients With Metastatic Renal Cell Carcinoma
Brief Title: A Clinical Study to Evaluate Safety and Immunologic Response of COMBIG-DC, in Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mendus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-101; 2011-002039-25 (EudraCT Number)
Record Dates: First submitted 2012-01-20; First posted 2012-02-02 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cancer Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combig-DC Cancer Vaccine (Experimental): Two vaccinations of Combig-DC (allogeneic dendritic cells) Cancer Vaccine given before nephrectomy.
  Interventions: Biological: Combig-DC (allogeneic dendritic cells) Cancer Vaccine

INTERVENTIONS:
Biological: Combig-DC (allogeneic dendritic cells) Cancer Vaccine — Cryopreserved dendritic cell suspension of 10 million cells per ml in heat-inactivated plasma, supplemented with 10% dimethyl sulfoxide (DMSO).

SUMMARY:
The primary objective of this study is to answer the question "Is it possible to inject the Combig-DC vaccine in a renal tumour without getting unacceptable side effects"? Patients newly diagnosed with metastatic renal cell carcinoma will get Combig-DC vaccinations at two occasions in a two weeks period (day 1 and day 14). After another two weeks the kidney will be eliminated. Adverse events will be registered, as well as changes in vital signs(heart rate, blood pressure and body temperature) and lab parameters. Immunologic response will be evaluated by measuring immunologic markers in blood and tumour tissue, and measuring the size of the metastases three months after nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Be informed of the nature of the study and have provided written informed consent
2. At least 18 years of age.
3. Diagnosis of renal cell carcinoma with at least one distant metastasis, and/or one distant lymph node metastasis.
4. Tumor size (renal cell carcinoma; primary tumor) at least 4.0 cm in longest diameter as measured by CT. Distant metastasis at least 1 cm diameter as measured by CT or a distant lymph node metastasis at least 2,5 cm diameter as measured by CT. Clinical stage 'T1b or more; NX; M1'
5. Adequate hematological parameters, i.e:

   B-Leukocyte count ≥ 4.5 x 109/L B-Platelet count ≥ 150 x109/L B-Haemoglobin ≥ 100 g/L
6. Women of Childbearing Potential (WOCBP) should use adequate contraception (oral or injectable contraceptives, hormone releasing intrauterine device) throughout the study period.

Exclusion Criteria:

1. Performance status > ECOG 2 after optimization of analgesics
2. Adequate coagulation parameters, i.e: P-Prothrombin complex (PK), P-APT time
3. Ongoing treatment with systemic corticosteroids (inhaled, intranasal and local steroids accepted) within 28 days before first vaccination.
4. Previously known or ongoing active autoimmune disease which requires treatment with systemic immunosuppressive agents. E.g. inflammatory bowel disease, multiple sclerosis, sarcoidosis, psoriasis, autoimmune hemolytic anemia, rheumatoid arthritis, SLE, vasculitis, Sjögren's syndrome, scleroderma, autoimmune hepatitis, and other rheumatological diseases.
5. Patients with previous or ongoing skin malignancy (basal-cell carcinoma, squamous cell carcinoma, melanoma), other hematological or solid malignancy or blood dysfunctions.
6. Ongoing infection that requires treatment with antibiotics.
7. Known major reaction/adverse event in connection with previously made vaccination (e.g. asthma, anaphylaxis or other serious reaction)
8. Known malignancy in CNS.
9. Active or latent virus disease (HIV, HBV and HCV).
10. Ongoing pregnancy or lactation. Females needs to have negative pregnancy test at screening visit.
11. Life expectancy less than 3 months.
12. Concomitant exposure to other investigational products.
13. Any reason that, in the opinion of the investigator, contraindicates that the patient participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Registration of adverse events as a measure of safety and tolerability | 1 year 3 months (Feb 2012-May 2013)
Changes in vital signs from baseline (heart rate, blood pressure, body temperature) as a measure of safety and tolerability | 1 year 3 months (Feb 2012 - May 2013)
Changes in lab parameters from baseline as a measure of safety and tolerability | 1 year 3 months (Feb 2012 - May 2013)

SECONDARY OUTCOMES:
Immunologic response in blood (immunologic panel) measured with ELISPOT. | 1 year 3 months (Feb 2012 - May 2013)
  Time for sampling: just before first injection and second injection, 2 weeks post second injection (in connection with the hospitalization for nephrectomy) and at 3 months post nephrectomy. ELISPOT assessment will be made at time of nephrectomy (after the second vaccination) at earliest.
Examination of immunohistology parameters (macrophage marker, CD3, CD4, CD8, CD56) of the renal tumor post nephrectomy. | 1 year 3 months (Feb 2012 - May 2013)
CT-evaluation of the size of the metastasis(-es) 3 months post nephrectomy | 1 year 3 months (Feb 2012 - March 2013)
CT evaluation to evaluate number of metastases 3 months post nephrectomy. | 1 year 3 months (Feb 2012 - May 2013)
Changes in body weight 3 months post nephrectomy vs. baseline. | 1 year 3 months (Feb 2012 - May 2013)
Changes in WHO-ECOG 3 months post nephrectomy vs. baseline. | 1 year 3 months (Feb 2012 - may 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Laurell, MD, PhD, Principal Investigator — Dept of Oncology , Uppsala University Hospital
Locations (1):
- Dept of Oncology, University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Laurell A, Lonnemark M, Brekkan E, Magnusson A, Tolf A, Wallgren AC, Andersson B, Adamson L, Kiessling R, Karlsson-Parra A. Intratumorally injected pro-inflammatory allogeneic dendritic cells as immune enhancers: a first-in-human study in unfavourable risk patients with metastatic renal cell carcinoma. J Immunother Cancer. 2017 Jun 20;5:52. doi: 10.1186/s40425-017-0255-0. eCollection 2017. PMID 28642820